CLINICAL TRIAL: NCT06023355
Title: Sex-related Differences in Outcome After Hybrid Coronary Revascularization Versus Coronary Artery Bypass Grafting in Multivessel Coronary Artery Disease: The SEX-HYBRID Study
Brief Title: Sex-related Differences in Outcome After Hybrid Coronary Revascularization
Acronym: SEX-HYBRID
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Associate Professor, University of Roma La Sapienza
Other Study IDs: 2023/D/1066
Record Dates: First submitted 2023-08-28; First posted 2023-09-05 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: HYBRID — It involves the combination of a sternal sparing left internal mammary artery (LIMA) bypass and percutaneous coronary intervention (PCI) with drug-eluting stents (DES) for non-left anterior descending (LAD) lesions. Through minimally invasive surgical techniques, HCR carries the potential for faster recovery postoperatively, fewer in-hospital complications, and lower utilization of healthcare resources, while providing the key benefits of LIMA-LAD grafting.

SUMMARY:
Hybrid coronary revascularization (HCR) has emerged as a favorable technique over traditional coronary artery bypass grafting (CABG) in a select group of patients with multivessel coronary artery disease (CAD). Till date, multiple individual studies comparing HCR with CABG have been carried out, but no data on the potential impact of sex on the outcome of HCR exist.

To fill this knowledge gap, the investigators aim to perform an international collaborative multi-center study in order to examine gender differences in short-term and long-term outcomes among patients who underwent HCR or CABG.

DETAILED DESCRIPTION:
Hybrid coronary revascularization (HCR) has emerged as a favorable technique over traditional coronary artery bypass grafting (CABG) in a select group of patients with multivessel coronary artery disease (CAD).

Till date, multiple individual studies comparing HCR with CABG have been carried out, but no data on the potential impact of sex on the outcome of HCR exist. Limited by their sample size, these individual studies may have been under-powered to detect a difference.

To fill this knowledge gap, the investigators aim to perform an international collaborative multi-center study in order to examine gender differences in short-term and long-term outcomes among patients who underwent HCR or CABG.

ELIGIBILITY:
Inclusion Criteria:

Patients with coronary artery disease and indication to cardiac surgery

Exclusion Criteria:

Contraindications to cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multivessel coronary artery disease and indication to cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Overall Mortality | Up to 1 year
  All causes deaths
Incidence of Composite End-point | Up to 1 year
  Cardiac death, myocardial infarction, stroke, bleeding

IPD SHARING:
Plan to Share IPD: Undecided